CLINICAL TRIAL: NCT07369375
Title: Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy and Safety of VMX Eye Drops for the Treatment of Dry Eye Disease (DED)
Brief Title: Efficacy and Safety of VMX Eye Drops for Dry Eye Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VISUfarma SpA (Industry)
Collaborators: CROlife (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMX-10-24
Record Dates: First submitted 2026-01-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group - VMX Eye Drops (Active Comparator)
  Interventions: Device: VMX Eye Drops
- Placebo Group - Placebo Eye Drops (Placebo Comparator)
  Interventions: Device: placebo eye drops

INTERVENTIONS:
Device: VMX Eye Drops — VMX ophthalmic solution; the dosage is one drop in each eye three times a day for 56 days.
  Arms: Treatment Group - VMX Eye Drops
Device: placebo eye drops — Sterile ophthalmic solution. The dosage is one drop in each eye three times a day for 56 days.
  Arms: Placebo Group - Placebo Eye Drops

SUMMARY:
This multicenter, randomized, double-blind study evaluates the safety and effectiveness of VMX eye drops in patients with dry eye disease. It aims to improve tear film stability, reduce dry eye symptoms, and enhance patients' quality of life compared to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an age of ≥ 18 and ≤ 80 years
* Patients with a diagnosis of Dry Eye (mild/moderate) with at least one of the following:

  * Tear Osmolarity >308 mOsm/L
  * TBUT < 10 seconds
  * Schirmer I test ≥ 5 mm and ≤ 14 mm at 5 minutes
* Patients not treated with artificial tears for at least 7 days
* Patients not treated with artificial tears for at least 7 days

Exclusion Criteria:

* Use of systemic medications which may affect a dry eye condition within 1 month prior to study enrolment (e.g. low-dose aspirin, antihistamines, decongestants, antipsychotics, parkinsonism medications, anticholinergics, oral isotretinoin, and oral diazepam)
* Patients with a score of ≤ 4 mm at 5 minutes on the Schirmer I test
* Patients that suffer of ocular allergy pathology (seasonal and chronic)
* Ongoing ocular or systemic infectious conditions
* Use of topical ocular therapies that cannot be suspended for the entire duration of the study
* Use of topical antibiotics and or corticosteroids within 15 days prior to study enrolment
* Use of systemic antibiotics and or corticosteroids within 1 month prior to study enrolment
* Any intraocular surgery in the past 12 months or require any intraocular surgery during the study
* Acute and Chronic Conjunctival Disease
* Eyelid surgery within the 6 months prior to study enrolment
* Presence of congenitally absent lacrimal or Meibomian glands or have any obstructive disease of the lacrimal glands
* History of ocular herpetic keratitis or active blepharitis in the 4 weeks prior to study enrolment
* History of autoimmune diseases
* Inflammations or abnormalities in the eyelid, in accordance with PI's clinical judgment
* History of corneal diseases, as keratoconus
* History of corneal transplant in one or both eyes
* Keratinization of the eyelid margin
* History of Sjögren's syndrome
* History of corneal trauma in the last 4 weeks prior to study enrolment
* Patients who are unwilling to discontinue all artificial tears and use only the study product ad indicated for the duration of the study
* Inability to self-administer study medications
* Women of childbearing potential who are pregnant, breast feeding, plan to become pregnant during the study, or not using adequate birth control methods to prevent pregnancy throughout the study.
* Any hypersensitivity to the use of the study product formulations or an allergy to any ingredients contained within product formulation
* Participation in other clinical studies involving drugs or devices within 30 days prior to study enrolment.
* Patients legally or mentally incapacitated unable to give informed consent for the participation in this trial
* Patients unable or unwilling to comply with appointments or all protocol requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Tear Break-up Time (TBUT) | From Baseline (V1) to Visit 3 (V3 - Day 56 after first administration)
  Assessment of the change in Tear Break-up Time (TBUT) at V3 versus V1 in the two groups.

SECONDARY OUTCOMES:
Tear Break-up Time (TBUT) | From Baseline (V1) to Visit 2 (V2 - Day 17 after first administration)
  Assessment of Tear Break-up Time (TBUT) at V2 compared to V1 in the two groups.
Schirmer I test | From Baseline (V1) to Visit 3 (V3 - Day 57 after first administration)
  Assessment of Schirmer I test at V2, and V3 compared to V1 in the two groups
Tear Osmolarity | From Baseline (V1) to Visit 3 (V3 - Day 57 after first administration)
  Assessment of Tear Osmolarity at V2, and V3 compared to V1 in the two groups
Ocular Surface Disease Index (OSDI) Questionnaire | From Baseline (V1) to Visit 3 (V3 - Day 57 after first administration)
  Assessment of Dry Eye symptoms at V1, V2 and V3, using the Ocular Surface Disease Index (OSDI) Questionnaire
Standard Patient Evaluation of Eye Dryness Questionnaire (SPEED) | From Baseline (V1) to Visit 3 (V3 - Day 57 after first administration)
  Assessment of Dry Eye symptoms at V1, V2 and V3, using Standard Patient Evaluation of Eye Dryness Questionnaire (SPEED)
Adverse Events | From first administration to Visit 3 (V3 - Day 57 after first administration)
  Quantitative and Qualitative Evaluation of Safety in terms of Adverse Events reported.

CONTACTS AND LOCATIONS:
Overall Officials: Anna R Bigioni, Study Chair — CROlife

IPD SHARING:
Plan to Share IPD: No